CLINICAL TRIAL: NCT06049680
Title: A Single-arm Open-label Safety Study of SMOFlipid to Evaluate the Risk of Developing Essential Fatty Acid Deficiency (EFAD) and/or Parenteral Nutrition-associated Cholestasis (PNAC) in Pediatric Patients 1 Month to 17 Years of Age and in Adult Patients, Who Are Anticipated to Need 8 Weeks or Longer of Parenteral Nutrition Treatment
Brief Title: Safety Study of SMOFlipid to Evaluate the Risk of Developing EFAD and/or PNAC in Pediatric and Adult Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMOF-044-CP4 (PMR 4240-1)
Record Dates: First submitted 2023-07-24; First posted 2023-09-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Malnutrition, Child; Malnutrition; Essential Fatty Acid Deficiency (EFAD); Parenteral Nutrition Associated Cholestasis
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — SMOFlipid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm SMOFlipid® (lipid injectable emulsion) (Other): Investigational drug: SMOFlipid® (lipid injectable emulsion).
  Interventions: Drug: SMOFlipid® (lipid injectable emulsion)

INTERVENTIONS:
Drug: SMOFlipid® (lipid injectable emulsion) — SMOFlipid is a sterile, nonpyrogenic, white, homogenous lipid emulsion for intravenous infusion. The lipid content of SMOFlipid is 0.20 g/mL, and comprises a mixture of soybean oil, MCT, olive oil, and fish oil. SMOFlipid belongs to the pharmacotherapeutic group: "Solutions for parenteral nutrition, fat emulsions" (ATC-code: B05BA02). SMOFlipid is indicated in adult and pediatric patients, including term and preterm neonates, as a source of calories and essential fatty acids for parenteral nutrition when oral or enteral nutrition is not possible, insufficient, or contraindicated.

SUMMARY:
Evaluate the risk of developing EFAD and/or PNAC in adult and pediatric patients 1 month of age and older, who are anticipated to need 8 weeks or longer of parenteral nutrition treatment with SMOFlipid.

ELIGIBILITY:
Age Limits: and Adults

Inclusion Criteria:

1. Male or female patients, at least 1 month of age.
2. Patients who require PN for at least 5 days/week.
3. Patients who receive 80% or more of their total energy requirements as PN at enrollment and who are expected to receive 80% or more of their total energy requirements as PN for at least 56 days.
4. Written informed consent. In case of pediatric patients, informed consent must be obtained from parent(s) or legal representatives. If possible, the assent of the pediatric patient must also be obtained (according to local law).

Exclusion Criteria:

1. Use of any other lipid injectable emulsion than SMOFlipid within 6 months prior to study participation
2. Known hypersensitivity to fish, egg, soybean, or peanut proteins, or to any of the active ingredients or excipients of SMOFlipid.
3. Hyperlipidemia or disorders of lipid metabolism characterized by hypertriglyceridemia (serum triglyceride concentration >250 mg/dL in infants or >400 mg/dL in older pediatric and adult patients).
4. Inborn errors of amino acid metabolism.
5. Cardiopulmonary instability (including pulmonary edema, cardiac insufficiency, myocardial infarction, acidosis and hemodynamic instability requiring significant vasopressor support).
6. Hemophagocytic syndrome.
7. Liver enzymes (either AST, or ALT, or GGT) exceeding 2 x upper limit of normal range
8. Direct bilirubin exceeding 2 x upper limit of normal range
9. INR exceeding 2 x upper limit of normal range and patient not receiving oral anticoagulants.
10. Any known hepatic condition outside of IFALD that will increase direct bilirubin ≥2.0 mg/dL.
11. Clinically significant abnormal levels of any serum electrolyte (sodium, potassium, magnesium, calcium, chloride, phosphate).
12. Active bloodstream infection demonstrated by positive blood culture at screening.
13. Severe renal failure (eGFR <15 ml/min per 1.73 m2) including patients on renal replacement therapy.
14. Abnormal blood pH, oxygen saturation, or carbon dioxide.
15. Pregnancy or lactation.
16. Participation in another interventional clinical study.
17. Unlikely to survive longer than 56 days.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of PNAC | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
  defined as direct bilirubin level > 2 mg/dL, confirmed by a second sample collected 7 days after the first sample
Time to direct bilirubin > 2mg/dL | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
  (confirmed by a second sample collected 7 days after the first)
Incidence of EFAD | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
  Triene/tetraene ratio in total plasma to assess EFAD (Holman 1960), Severity of EFAD will be graded based on triene/tetraene ratio, as suspected ≥ 0.05, moderate ≥ 0.20 and severe ≥ 0.40 (Cober et al 2012)
Incidence of clinical EFAD | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Fatty acids | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
  analyzed in total plasma, including linoleic acid, α-linolenic acid, arachidonic acid, docosahexaenoic acid, eicosapentaenoic acid and Mead acid

SECONDARY OUTCOMES:
Laboratory values: triglycerides | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: direct bilirubin | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: total bilirubin | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: alanine aminotransferase (ALT) | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: aspartate aminotransferase (AST) | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: gamma-glutamyl transferase (GGT) | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: alkaline phosphatase (ALP) | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: creatinine | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: urea nitrogen | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: electrolytes | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: glucose | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values: total protein | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values hematology: white blood cell count (WBC), red blood cell count (RBC), and platelet count | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values hematology: Hemoglobin | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values hematology Hematocrit | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Laboratory values hematology: International normalized ratio | At baseline before start of treatment to assess eligibility
Vital signs: Blood pressure | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Vital signs: Heart rate | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Vital signs: Body temperature | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
Incidence of adverse events | Start of Treatment until After End of Last Study PN (+6 months for pediatric patients). Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
BMI | Start of Treatment until After End of Last Study PN Duration of Treatment: Study treatment will last for a minimum of 8 weeks (56 consecutive days) and as long as PN is indicated, up to 1 year (365 consecutive days).
  BMI is the weight in kilograms divided by height in meters squared. Alternatively, BMI can be calculated by dividing the weight in kilograms by the height in centimeters squared, and then multiplying the result by 10,000.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rudolph, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Emory University Hospital, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania